CLINICAL TRIAL: NCT02452242
Title: A Phase 2, Dose Escalation, Schedule Comparison Study to Evaluate the Safety, Pharmacokinetics, and Viral Kinetics of ABX464 in Untreated Patients With HIV Infection in Mauritius
Brief Title: Safety, PK and PD Study of ABX464 in Untreated HIV Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Abivax S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ABX464-003
Record Dates: First submitted 2015-04-10; First posted 2015-05-22 (Estimated); Last update posted 2016-05-30 (Estimated); Status verified 2015-05

CONDITIONS: Human Immunodeficiency Virus Infections
MeSH Terms: interventions — ABX464

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ABX464 (Experimental)
  Interventions: Drug: ABX464
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: ABX464 — 25, 50, 75, 100, 150 mg, i.e. 1, 2, 3, 4 or 6 capsules respectively, every 3 days or every day for 2 weeks
  Arms: ABX464
Other: Placebo — 1, 2, 3, 4 or 6 capsules respectively, every 3 days or every day for 2 weeks
  Arms: Placebo

SUMMARY:
ABX464 is a first in class that showed efficacy as an anti-HIV therapy. The present study is intended to assess the safety, the tolerability, and pharmacokinetic parameters and to evaluate the effect on viral load of repeated oral administrations of ABX464 in patients infected by HIV, not previously treated for their HIV.

Two types of design are intended in this protocol: dosing every 3 days or dosing every day. The goal is to determine the best dosing regimen to reduce viral load and minimize adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females, 18 to 65 years of age
2. Patients infected by HIV-1 or HIV-2
3. BMI between 17 and 29 kg/m².
4. CD4 cell count ≥ 350 /mm3 and HIV RNA level between 5,000-500,000 copies/mL.
5. Clinical laboratory tests (hematology, blood chemistry, and urinalyses) must be within normal limits, or clinically acceptable to the sponsor and principal investigator and consistent with the underlying HIV infection.
6. Urine drug screen for drugs with a high potential for abuse (cocaine, opiates, amphetamines and barbiturates) and alcohol breath test must be negative.
7. Females must be non lactating and either be of nonchildbearing potential (ie sterilized via hysterectomy or bilateral tubal ligation or at least one year post-menopausal) or if of child bearing potential, must be practicing effective double barrier contraceptive methods from at least two weeks prior to Day 1 until 3 months after the last dose of study medication.
8. Males must practice an effective barrier method of contraception from Day 1 until 3 months days after the last dose of study medication.
9. Patients must be willing to give written informed consent prior to study enrollment and be able to adhere to restrictions and examination schedules.
10. Physical examination and ECG must be within normal limits.
11. Never taken any antiretroviral agent except for a brief time, and for some reasons, the patient decided not to continue therapy (i.e. Toxicity, personal decision. None in past 30-180 days.

Exclusion Criteria:

1. Individuals with a history of any significant medical disorders which requires a physician's care.
2. Individuals who have a history of any clinically significant local or systemic infectious disease (other than HIV-1 or HIV-2 infection) within four weeks prior to drug administration.
3. Individuals with any clinically significant laboratory abnormalities as defined as grade 2 or 3 in Common Terminology Criteria for Adverse Events (CTCAE), version 4.0.
4. Individuals who are positive for hepatitis B virus and/or hepatitis C virus
5. Any individual who does not comply with the requirement that he should not have used any drugs (including prescription, nonprescription, herbal, and mineral supplements) other than paracetamol for at least two weeks prior to the study nor alcohol within 48 hours prior to drug administration and for the entire study period. The use of a concomitant medications to treat an AE during the study will not be considered a protocol violation.
6. Individuals who have participated in a clinical trial of an investigational drug within 90 days prior to the start of the study
7. Individuals who smoke more than ten cigarettes or equivalent tobacco use per day.
8. Individuals with forfeiture of freedom by an administrative or legal obligation or under guardianship

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2015-01; Primary Completion 2015-12 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability profile of ABX464 as assessed by the change from baseline in laboratory values, in vital signs and ECG parameters at week 3 and by the number of patients with adverse events. | Week 3
  Number of patients with abnormal blood (hematology and biochemistry) and urinary laboratory values, abnormal vital signs and ECG parameters and the number/proportion of patients reporting any adverse event.

SECONDARY OUTCOMES:
Cmax | week 1, week 2 and week 3
  Maximum concentration in plasma of ABX464 and metabolite
tmax | Week 3
  Time to maximum concentration
AUC | Week 3
  Area under the concentration-time curve
t1/2 | Week 3
  Half-life of the ABX464 in plasma
Pharmacodynamic activity as expressed by CD4 and CD8 count | Week 3
  CD4 and CD8 values
Pharmacodynamic activity as expressed by HIV viral load | Week 3
  HIV viral load across time and possible relationship with PK parameters

CONTACTS AND LOCATIONS:
Locations (4):
- CAP Research Ltd, Curepipe, Mauritius
- Thailand (3):
  - HIV-NAT, Thai Red Cross AIDS Research Center, Bangkok
  - Siriraj Hospital, Mahidol University, Bangkok
  - Chiang Mai University, Chiang Mai

REFERENCES:
- [Derived] Steens JM, Scherrer D, Gineste P, Barrett PN, Khuanchai S, Winai R, Ruxrungtham K, Tazi J, Murphy R, Ehrlich H. Safety, Pharmacokinetics, and Antiviral Activity of a Novel HIV Antiviral, ABX464, in Treatment-Naive HIV-Infected Subjects in a Phase 2 Randomized, Controlled Study. Antimicrob Agents Chemother. 2017 Jun 27;61(7):e00545-17. doi: 10.1128/AAC.00545-17. Print 2017 Jul. PMID 28507108